CLINICAL TRIAL: NCT01042704
Title: Phase I Study of Bendamustine in Combination With Lenalidomide (CC-5013) and Dexamethasone in Patients With Refractory or Relapsed Multiple Myeloma
Brief Title: Bendamustine in Combination With Lenalidomide and Dexamethasone in Refractory or Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Redner, MD (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor-Investigator, Robert Redner, MD, Professor, Division of Hematology/Oncology, Department of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-089
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Myeloma
Keywords: Relapsed Myeloma; Refractory Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Bendamustine Hydrochloride; Lenalidomide; Dexamethasone; Aspirin; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine, Lenalidomide and Dexamethasone (Experimental): Treatment with Bendamustine in combination with Lenalidomide and Dexamethasone will be administered on an outpatient basis. Each treatment cycle will be 28 days dosed according to the Dose Escalation Schema.
  Interventions: Drug: Bendamustine; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Aspirin; Drug: Prophylaxis; Drug: Antibiotic; Other: Biweekly Follow Up; Other: Cyclical Follow Up; Other: Restaging; Other: Post-Treatment Follow Up

INTERVENTIONS:
Drug: Bendamustine — Bendamustine is given intravenously (into a vein or IV infusion) on days 1 and 2 of each cycle. Each bendamustine infusion will take 60 minutes
Drug: Lenalidomide — Lenalidomide is taken orally (by mouth) in the morning on days 1 through 21 of each cycle.
Drug: Dexamethasone — Dexamethasone is taken orally (by mouth) on days 1, 8, 15, and 22 of each cycle.
Drug: Aspirin — All patients will receive enteric coated aspirin, 325 mg, QD while on study. If patient is unable to tolerate aspirin, patient should receive other types of anti-coagulation like Coumadin or low molecular weight heparin.
Drug: Prophylaxis — All patients will receive prophylaxis with either an H-2 blocker or proton pump inhibitor (PPI) while on study medications. Suggested medications included ranitidine 150 mg PC BID or omeprazole 20 mg PO QD or equivalent.
Drug: Antibiotic — PCP antibiotic prophylaxis with a Bactrim will be recommended. In case of history of zoster or fungal infection a prophylaxis with Acyclovir or Diflucan should be also considered.
Other: Biweekly Follow Up — Vital signs (heart rate, breathing rate, blood pressure, and temperature) will be measured, and Blood tests to check CBC, Calcium, Electrolytes, serum, creatinine, and BUN. This follow up will take place at the Hillman Cancer Center, or whichever cancer center in which the subject is treated.
Other: Cyclical Follow Up — At the beginning of each treatment cycle subjects will undergo a Physical exam, a Performance status check, Recording of any new symptoms or side effects and any new medications, Blood tests (including blood chemistry, organ function and indicators of disease), Urine test, and pregnancy test (if applicable).
Other: Restaging — Every other cycle subjects' disease will be restaged. This will be accomplished by their treatment physician. Re-staging procedures includes a regular office visit, x-ray, and a bone marrow biopsy. Subjects will spend approximately 4 hours at the Hillman Cancer Center or the UPMC Cancer Center location where they are being treated for this re-staging.
Other: Post-Treatment Follow Up — After subjects stop receiving the study drugs, they will be followed every 3 months for the first two years, every 6 months for years 2-5, and annually thereafter. The following procedures, which are considered routine for their cancer care, will be done as part of this follow-up:
  * Physical exam
  * Performance status (check of ability to perform daily functions)
  * Recording of any new symptoms and any new medications being taken
  * Blood tests to check blood counts (numbers of red and white blood cells and platelets), blood chemistry (to check organ function), and indicators of disease (immunoglobulins)
  * Urine test (24hr urine)
  * Women who are able to have children will have a pregnancy test (4 weeks after their last dose of lenalidomide).
  * A check of the status of disease (includes bone marrow biopsy, skeletal survey, and blood and urine tests). Bone marrow biopsy will be done at the end of treatment, if subjects have a complete response, and their disease gets worse.

SUMMARY:
The purpose of this study is to see if the combination of bendamustine, lenalidomide and dexamethasone will help people with multiple myeloma that has returned after standard treatment or has been resistant to other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed symptomatic Multiple Myeloma, Salmon-Durie Stage II or III or International Staging System II or III that has been previously treated with at least one cycle of a specific therapy; after which the patient has shown progressive or refractory disease, and must meet at least one of the following parameters of measurable disease:
* Bone marrow plasmacytosis with > 10% plasma cells, or sheets of plasma cells, or biopsy proven plasmacytoma which must be obtained within 6 weeks prior to registration.
* Measurable levels of monoclonal protein (M protein): > 1 g/dL of IgG or IgM M-protein or > 0.5 g/dL IgA or IgD M protein on serum protein electrophoresis OR > 200 mg of free light chain on a 24 hour urine protein electrophoresis which must be obtained within 4 weeks prior to registration OR > 20 mg/dL involved free light chain on serum free light chain testing with an abnormal kappa:lambda light chain ratio. Note that if both serum and urine m-components are present, both must be followed in order to evaluate response. Both SPEP and UPEP must be performed within 28 days prior to registration.
* Patients with lytic bone disease, defined as at least one lytic lesion that can be accurately measured in at least one dimension.
* Patients must have received prior chemotherapy for their myeloma, but not in the last 4 weeks. Patients may have previously received autologous peripheral blood stem cell transplantation. Prior treatment with lenalidomide is allowed.
* Patients should not have received any radiation for the preceding 4 weeks before entry onto the study. Exception: local radiation therapy for symptomatic bone lesions (eg,uncontrolled pain or high risk of pathologic fracture)
* Age >= 18 years
* Life expectancy of greater than 6 months.
* ECOG performance status >=2 (Karnofsky >=60%). Patients with PS of 3 are eligible if their PS is due to pain, which would likely improve with treatment.
* Patients must have normal organ and marrow function as defined below, obtained within 4 weeks prior to registration:

  * Hgb > 9 g/dL (which may be supported by transfusion or growth factors)
  * leukocytes >=2,000/ml
  * absolute neutrophil count ≥1000/ ml
  * platelets >=75,000/mcL
  * total bilirubin >=2.5 mg/dl
  * AST(SGOT)/ALT(SGPT) >=5 X institutional upper limit of normal
  * creatinine <2.5 mg/dl
* Patients must not be pregnant or breast feeding. Due to the potential teratogenic properties of lenalidomide, the use of this drug in patients that are pregnant is absolutely contraindicated. Further, all women of childbearing potential and sexually active males must agree to avoid conception while participating in this study. Specifically, women of childbearing potential must either agree to refrain from sexual intercourse or employ a dual method of contraception, one of which is highly effective (IUD, birth control pills, tubal ligation or partners vasectomy), and another additional method (condom, diaphragm, or cervical cap) for 4 weeks prior to receiving lenalidomide, and for four weeks after discontinuing this therapy. Sexually active males cannot participate unless they agree to use a condom (even if they have undergone a prior vasectomy) while having intercourse with a woman of child bearing potential while taking lenalidomide and for four weeks after stopping treatment. Women of child bearing potential (those who have not had a hysterectomy or the absence of menstrual periods for at least 24 consecutive months) must have a negative pregnancy test 10-14 days prior to the initiation of therapy and a repeat negative pregnancy test 24 hours prior to the initiation of lenalidomide.
* Ability to understand and the willingness to sign a written informed consent document. Patient must be informed of the investigational nature of this study.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Exception: local radiation therapy for symptomatic bone lesions (eg, uncontrolled pain or high risk of pathologic fracture)
* Patients receiving any other investigational agents.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide and/or Bendamustine or other agents used in the study.
* Patients with a second malignancy other than squamous/basal cell carcinoma of the skin or in situ carcinoma of the cervix unless the tumor was curatively treated at least two years previously.
* Inability to comply with study and/or follow-up procedures.
* If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:

  * Must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices).
  * Must have a platelet count >75,000.
  * Must have stable INR between 2-3.
* Patients who have not collected hematopoietic progenitors and are potential candidates for autologous transplantation .
* Patients that have a serious cardiac condition, such as myocardial infarction within 6 months or heart disease as defined by the New York Heart Association Class III or IV,
* Patients with prior allogeneic stem cell transplant.
* Non-secretory patients (i.e., patients who do not meet the minimum M-protein or light chain criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To establish the dose of each drug recommended for a future Phase II protocol with the combination | 1 year

SECONDARY OUTCOMES:
To explore anti-tumor activity of the combination of Bendamustine plus Lenalidomide and dexamethasone | 2.5 years
Toxicity, time to progression, overall survival. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Redner, M.D., Principal Investigator — University of Pittsburgh Physicians, Hematology/Oncology
Locations (22):
- United States (22):
  - Karmanos Cancer Institute, Detroit, Michigan
  - UPMC Cancer Centers - Teramana Cancer Center, Steubenville, Ohio
  - UPMC Cancer Centers - Beaver, Beaver, Pennsylvania
  - UPMC Cancer Centers - Jefferson, Clairton, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer at Mountain View, Greensburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer at Oakbrook, Greensburg, Pennsylvania
  - UPMC Cancer Centers - Indiana, Indiana, Pennsylvania
  - UPMC Cancer Centers - Johnstown, Johnstown, Pennsylvania
  - Hematology-Oncology Associates of UPCI, McKeesport, Pennsylvania
  - Hematology/Oncology - Private Practice, McKeesport, Pennsylvania
  - UPMC Cancer Centers - Monroeville, Monroeville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer at Mt. Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Cancer Centers - New Castle, New Castle, Pennsylvania
  - UPMC Cancer Centers - St. Margaret's, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers - Passavant, Pittsburgh, Pennsylvania
  - VA Healthcare System - 646, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers - Drake, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers - Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Centers - Washington, Washington, Pennsylvania
  - UPMC Cancer Centers - North Hills, Wexford, Pennsylvania
  - UPMC Cancer Centers - Windber, Windber, Pennsylvania

REFERENCES:
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Londono F. Thalidomide in the treatment of actinic prurigo. Int J Dermatol. 1973 Sep-Oct;12(5):326-8. doi: 10.1111/j.1365-4362.1973.tb00066.x. No abstract available. PMID 4747626
- [Background] Vogelsang GB, Farmer ER, Hess AD, Altamonte V, Beschorner WE, Jabs DA, Corio RL, Levin LS, Colvin OM, Wingard JR, et al. Thalidomide for the treatment of chronic graft-versus-host disease. N Engl J Med. 1992 Apr 16;326(16):1055-8. doi: 10.1056/NEJM199204163261604. PMID 1549151
- [Background] Hayashi T, Hideshima T, Akiyama M, Podar K, Yasui H, Raje N, Kumar S, Chauhan D, Treon SP, Richardson P, Anderson KC. Molecular mechanisms whereby immunomodulatory drugs activate natural killer cells: clinical application. Br J Haematol. 2005 Jan;128(2):192-203. doi: 10.1111/j.1365-2141.2004.05286.x. PMID 15638853
- [Background] Strasser K, Ludwig H. Thalidomide treatment in multiple myeloma. Blood Rev. 2002 Dec;16(4):207-15. doi: 10.1016/s0268-960x(02)00031-0. PMID 12350364
- [Background] Tohnya TM, Figg WD. Immunomodulation of multiple myeloma. Cancer Biol Ther. 2004 Nov;3(11):1060-1. doi: 10.4161/cbt.3.11.1303. Epub 2004 Nov 12. PMID 15640623
- [Background] Lentzsch S, LeBlanc R, Podar K, Davies F, Lin B, Hideshima T, Catley L, Stirling DI, Anderson KC. Immunomodulatory analogs of thalidomide inhibit growth of Hs Sultan cells and angiogenesis in vivo. Leukemia. 2003 Jan;17(1):41-4. doi: 10.1038/sj.leu.2402745. PMID 12529658
- [Background] Singhal S, Mehta J, Desikan R, Ayers D, Roberson P, Eddlemon P, Munshi N, Anaissie E, Wilson C, Dhodapkar M, Zeddis J, Barlogie B. Antitumor activity of thalidomide in refractory multiple myeloma. N Engl J Med. 1999 Nov 18;341(21):1565-71. doi: 10.1056/NEJM199911183412102. PMID 10564685
- [Background] Anagnostopoulos A, Weber D, Rankin K, Delasalle K, Alexanian R. Thalidomide and dexamethasone for resistant multiple myeloma. Br J Haematol. 2003 Jun;121(5):768-71. doi: 10.1046/j.1365-2141.2003.04345.x. PMID 12780791
- [Background] Podar K, Anderson KC. The pathophysiologic role of VEGF in hematologic malignancies: therapeutic implications. Blood. 2005 Feb 15;105(4):1383-95. doi: 10.1182/blood-2004-07-2909. Epub 2004 Oct 7. PMID 15471951
- [Background] Palumbo A, Bertola A, Musto P, Caravita T, Callea V, Nunzi M, Grasso M, Falco P, Cangialosi C, Boccadoro M. Oral melphalan, prednisone, and thalidomide for newly diagnosed patients with myeloma. Cancer. 2005 Oct 1;104(7):1428-33. doi: 10.1002/cncr.21342. PMID 16116606
- [Background] Richardson PG, Schlossman RL, Weller E, Hideshima T, Mitsiades C, Davies F, LeBlanc R, Catley LP, Doss D, Kelly K, McKenney M, Mechlowicz J, Freeman A, Deocampo R, Rich R, Ryoo JJ, Chauhan D, Balinski K, Zeldis J, Anderson KC. Immunomodulatory drug CC-5013 overcomes drug resistance and is well tolerated in patients with relapsed multiple myeloma. Blood. 2002 Nov 1;100(9):3063-7. doi: 10.1182/blood-2002-03-0996. PMID 12384400
- [Background] Zangari M, Tricot G, Zeldis J, Eddlemon P, Saghafifar F, Barlogie B. Results of phase I study of CC-5013 for the treatment of multiple myeloma (MM) patients who relapse after high dose chemotherapy (HDCT). Blood. 2001 :775a (A3226).
- [Background] Richardson P, Jagannath 5, Schlossman R, eta!. A multi-center, randomized, phase 2 study to evaluate the efficacy and safety of 2 CC-5013 dose regimens when used alone or in combination with dexamethasone (Dex) for the treatment of relapsed or refractory multiple myeloma (MM). Blood. 2003;1 02:235a.
- [Background] Davies FE, Raje N, Hideshima T, Lentzsch S, Young G, Tai YT, Lin B, Podar K, Gupta D, Chauhan D, Treon SP, Richardson PG, Schlossman RL, Morgan GJ, Muller GW, Stirling DI, Anderson KC. Thalidomide and immunomodulatory derivatives augment natural killer cell cytotoxicity in multiple myeloma. Blood. 2001 Jul 1;98(1):210-6. doi: 10.1182/blood.v98.1.210. PMID 11418482
- [Background] Hideshima T, Chauhan D, Podar K, Schlossman RL, Richardson P, Anderson KC. Novel therapies targeting the myeloma cell and its bone marrow microenvironment. Semin Oncol. 2001 Dec;28(6):607-12. doi: 10.1016/s0093-7754(01)90033-8. PMID 11740818
- [Background] Hideshima T, Chauhan D, Shima Y, Raje N, Davies FE, Tai YT, Treon SP, Lin B, Schlossman RL, Richardson P, Muller G, Stirling DI, Anderson KC. Thalidomide and its analogs overcome drug resistance of human multiple myeloma cells to conventional therapy. Blood. 2000 Nov 1;96(9):2943-50. PMID 11049970
- [Background] Mitsiades N, Mitsiades CS, Poulaki V, Chauhan D, Richardson PG, Hideshima T, Munshi NC, Treon SP, Anderson KC. Apoptotic signaling induced by immunomodulatory thalidomide analogs in human multiple myeloma cells: therapeutic implications. Blood. 2002 Jun 15;99(12):4525-30. doi: 10.1182/blood.v99.12.4525. PMID 12036884
- [Background] Dimopoulos MA, Spencer A, Attal M, a!. e. Study of lenalidomide plus dexamethasone versus dexamethasone alone in relapsed or refractory multiple myeloma (MM); results of a phase 3 study (MM-01 0). Blood. 2005:106:1 06a (abstract).
- [Background] Weber DM, Chen D, Niesvizky R, et al. Lenalidomide plus high-dose dexamethasone provides improved overall survival compared to high-dose dexamethasone alone for relapsed or refractory multiple myeloma (MM): results of a North American phase Ill study (MM-009). Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings. 2006;24(1 8S):Abstract #7521.
- [Background] Schrijvers D, Vermorken JB. Phase I studies with bendamustine: an update. Semin Oncol. 2002 Aug;29(4 Suppl 13):15-8. doi: 10.1053/sonc.2002.34874. PMID 12170427
- [Background] Ponisch W, Mitrou PS, Merkle K, Herold M, Assmann M, Wilhelm G, Dachselt K, Richter P, Schirmer V, Schulze A, Subert R, Harksel B, Grobe N, Stelzer E, Schulze M, Bittrich A, Freund M, Pasold R, Friedrich T, Helbig W, Niederwieser D; East German Study Group of Hematology and Oncology (OSHO). Treatment of bendamustine and prednisone in patients with newly diagnosed multiple myeloma results in superior complete response rate, prolonged time to treatment failure and improved quality of life compared to treatment with melphalan and prednisone--a randomized phase III study of the East German Study Group of Hematology and Oncology (OSHO). J Cancer Res Clin Oncol. 2006 Apr;132(4):205-12. doi: 10.1007/s00432-005-0074-4. Epub 2006 Jan 10. PMID 16402269
- [Background] Ponisch W, Rozanski M, Goldschmidt H, Hoffmann FA, Boldt T, Schwarzer A, Ritter U, Rohrberg R, Schwalbe E, Uhlig J, Zehrfeld T, Schirmer V, Haas A, Kreibich U, Niederwieser D; East German Study Group of Haematology and Oncology (OSHO). Combined bendamustine, prednisolone and thalidomide for refractory or relapsed multiple myeloma after autologous stem-cell transplantation or conventional chemotherapy: results of a Phase I clinical trial. Br J Haematol. 2008 Oct;143(2):191-200. doi: 10.1111/j.1365-2141.2008.07076.x. Epub 2008 Aug 24. PMID 18752593
- [Background] Balfour JA, Goa KL. Bendamustine. Drugs. 2001;61(5):631-8; discussion 639-40. doi: 10.2165/00003495-200161050-00009. PMID 11368287
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Hrusovsky I, Heidtmann H, (ASH Annual Meeting Abstracts) Blood 2005 106:abstract 5122
- [Derived] Lentzsch S, O'Sullivan A, Kennedy RC, Abbas M, Dai L, Pregja SL, Burt S, Boyiadzis M, Roodman GD, Mapara MY, Agha M, Waas J, Shuai Y, Normolle D, Zonder JA. Combination of bendamustine, lenalidomide, and dexamethasone (BLD) in patients with relapsed or refractory multiple myeloma is feasible and highly effective: results of phase 1/2 open-label, dose escalation study. Blood. 2012 May 17;119(20):4608-13. doi: 10.1182/blood-2011-12-395715. Epub 2012 Mar 26. PMID 22451423